CLINICAL TRIAL: NCT06209047
Title: A Randomized Sham-Controlled Trial of Bronchoscopic Levofloxacin and Gentamicin Versus Sham in Mechanically Ventilated Bronchiectasis: Acute and 1-Year Outcomes
Brief Title: Bronchoscopic Levofloxacin, Gentamicin, or Sham for Acute Exacerbation of Bronchiectasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Abuzaid Ali, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AU-12578383
Record Dates: First submitted 2023-12-26; First posted 2024-01-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Bronchiectasis With Acute Exacerbation
Keywords: Bronchiectasis; Bronchoscopy; Levofloxacin; Gentamicins; Steroids
MeSH Terms: conditions — Bronchiectasis | interventions — Budesonide; Steroids; Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: Arm 1: Levofloxacin
  Bronchoscopic instillation of levofloxacin 500 mg in isotonic saline during standardized bronchoscopy.
  Arm 2: Gentamicin
  Bronchoscopic instillation of gentamicin 80 mg in isotonic saline during standardized bronchoscopy.
  Arm 3: Sham
  Bronchoscopy for airway visualization only, no lavage or drug instillation (sham procedure).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) All participants, clinical care providers (including bedside staff), investigators, and outcomes assessors will be blinded to group allocation. The use of a sham bronchoscopic procedure in the control arm ensures that all patients undergo a procedure of similar appearance and duration, minimizing the risk of performance and detection bias. Unblinding will only occur in the event of medically necessary interventions during the sham procedure, which will be documented as protocol deviations while maintaining the intention-to-treat analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gentamicin group (Experimental): This arm will undergo bronchoscopic airway clearance followed by local instillation of gentamicin (80 mg once) and Budesonide (0.5 mg) once.
  Interventions: Drug: Local instillation of gentamicin and Budesonide; Procedure: Bronchoscopic mechanical secretion suction and lavage
- Levofloxacin group (Experimental): This arm will undergo bronchoscopic airway clearance followed by bronchoscopic instillation of levofloxacin 480 mg in isotonic saline during standardized bronchoscopy. And Budesonide (0.5 mg) once.
  Interventions: Drug: Local instillation of Levofloxacin and Budesonide; Procedure: Bronchoscopic mechanical secretion suction and lavage
- Sham group (Sham Comparator): Bronchoscopy for airway visualization only, no lavage or drug instillation (sham procedure).
  Interventions: Procedure: Sham Bronchoscopy

INTERVENTIONS:
Drug: Local instillation of gentamicin and Budesonide — Bronchoscopic local instillation of gentamicin and Budesonide
  Other Names: Bronchoscopic instillation of gentamicin and steroids
  Arms: Gentamicin group
Drug: Local instillation of Levofloxacin and Budesonide — Bronchoscopic local instillation of Levofloxacin and Budesonide
  Other Names: Bronchoscopic instillation of levofloxacin and steroids
  Arms: Levofloxacin group
Procedure: Bronchoscopic mechanical secretion suction and lavage — Bronchoscopic mechanical secretion suction and lavage
  Arms: Gentamicin group; Levofloxacin group
Procedure: Sham Bronchoscopy — Bronchoscopy for airway visualization only, no lavage or drug instillation (sham procedure).
  Other Names: Masking intervention
  Arms: Sham group

SUMMARY:
Randomized single-center trial evaluating whether bronchoscopic instillation of levofloxacin or gentamicin improves outcomes compared to a sham bronchoscopic procedure in adult ICU patients with non-cystic fibrosis bronchiectasis requiring invasive mechanical ventilation. The primary outcome is a ranked composite of in-hospital mortality and time to ventilator liberation. Safety and procedural adverse events are closely monitored.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic suppurative and inflammatory lung disease of diverse etiology characterized by pathological and irreversible dilatation of the bronchial tree. The impairment of the mucociliary clearance, which results from chronic airway inflammation, may cause long-term colonization or recurrent infection of bacteria, especially Pseudomonas aeruginosa (PA), while bacterial colonization and recurrent infection can aggravate airway inflammation. Sputum retention caused by the impairment of mucociliary clearance can result in mucous plugs, which in turn contribute to airflow obstruction and dyspnea.

Clinically, the major manifestations of bronchiectasis include chronic cough with purulent sputum, dyspnea, and fatigue, which can significantly diminish patients' quality of life. The frequency of exacerbations and decline in lung function may lead to a poor prognosis and a decrease in quality of life.

The purpose of bronchiectasis management is to reduce exacerbations, prevent complications, and improve the quality of life. Long-term instillation of antibiotics and steroids can reduce the concentration of bacteria in the airways, decrease sputum production, attenuate lung function decline, and reduce acute pulmonary exacerbations without nephrotoxicity or ototoxicity. Dexamethasone is one of the most common glucocorticoids that can inhibit the expression levels of inflammatory factors in the airway and reduce the secretion of airway mucus. Topical administration could also reduce the systemic side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients with bronchiectasis confirmed by high-resolution CT chest(HRCT)
* patients with acute exacerbation of bronchiectasis who need antibiotic treatment at the hospital due to exacerbation
* mechanically ventilated patients in the respiratory ICU
* Age more than or equal to 18 years

Exclusion Criteria:

* patients with active pulmonary tuberculosis
* patients with allergic bronchopulmonary aspergillosis
* patients who underwent interventional bronchoscopy for hemoptysis
* age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Days for weaning from mechanical ventilation | one month
  days of mechanical ventilation will be measured and compared between drug and conventional groups

SECONDARY OUTCOMES:
The amount of sputum production per day(ml/day) | one year
  The total amount of sputum per day will be measured and compared between the drug and conventional groups
6-minute walking distance (meters) | one year
  The total recorded distance in 6 minutes in meters
number of exacerbations (recorded number/year) | one year
  The number of reported exacerbations in one year
Hospital admission | one year
  The number of reported hospital admissions in one year
Quality of life assessment in bronchiectasis patients | one year
  The quality of life assessment in bronchiectasis patients using patient-reported outcome measures (Quality of Life Bronchiectasis questionnaire). It consists of 8 domains scored on a 0 - 100 scale (higher equals better QoL)
Evaluation of anxiety in bronchiectasis patients using the Hamilton Anxiety rating Scale | one year
  The anxiety in bronchiectasis patients will be measured using the Hamilton Anxiety rating scale, which consists of 14 items ranging from 0 - 56 (higher equals more anxiety).
Evaluation of depression in bronchiectasis patients using the Hamilton Depression Rating Scale | one year
  The depression in bronchiectasis patients will be measured using the Hamilton Depression rating scale, which consists of 17 items ranging from 0 - 52 (higher equals more depression).

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Ali, MSc, Principal Investigator — Assiut University; Aliae A Hussien, MD, Study Chair — Assiut University; Ahmad M Shaddad, MD, Study Director — Assiut University; Maiada K Hashem, MD, Study Director — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All participant data will be recorded using a unique, study-specific Participant Identification (PID) number. This PID is not derived from any personal information and will be used for all data collection, analysis, and future data sharing. All datasets intended for sharing or publication will be thoroughly de-identified, with no direct or indirect personal identifiers included.
  Results from this trial will be published in two main peer-reviewed manuscripts: one reporting outcomes from the acute hospitalization phase (primary analysis), and a second reporting on long-term, 1-year follow-up outcomes. Both publications will use only de-identified PID-linked data and will cite the same ClinicalTrials.gov registration number.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 12 months after publication of the primary (acute phase) results, for a period of 3 years.
  Data from both the acute hospital phase and the 1-year follow-up phase will be available after publication of the respective results in peer-reviewed journals.
Access Criteria: De-identified individual participant data (IPD) will be made available to qualified researchers following publication of the primary and long-term results. Access will be granted for methodologically sound proposals that are consistent with the approved protocol and ethical standards. All requests must include a clear scientific rationale, analysis plan, and evidence of appropriate institutional review board (IRB) approval or waiver.
  Data will be shared under a data use agreement, which ensures:
  No attempt to re-identify participants, Use of data only for the approved research purpose, Compliance with all applicable privacy and security regulations. Requests will be reviewed by the trial's Steering Committee and Data Access Committee. Approved researchers will receive de-identified, PID-linked datasets and supporting documentation.
  To request data access, interested parties should contact the Principal Investigator.

REFERENCES:
- [Result] Chan SC, Shum DK, Tipoe GL, Mak JC, Leung ET, Ip MS. Upregulation of ICAM-1 expression in bronchial epithelial cells by airway secretions in bronchiectasis. Respir Med. 2008 Feb;102(2):287-98. doi: 10.1016/j.rmed.2007.08.013. Epub 2007 Oct 10. PMID 17931847
- [Result] Murray MP, Govan JR, Doherty CJ, Simpson AJ, Wilkinson TS, Chalmers JD, Greening AP, Haslett C, Hill AT. A randomized controlled trial of nebulized gentamicin in non-cystic fibrosis bronchiectasis. Am J Respir Crit Care Med. 2011 Feb 15;183(4):491-9. doi: 10.1164/rccm.201005-0756OC. Epub 2010 Sep 24. PMID 20870753
- [Result] King PT, Holdsworth SR, Freezer NJ, Villanueva E, Holmes PW. Characterisation of the onset and presenting clinical features of adult bronchiectasis. Respir Med. 2006 Dec;100(12):2183-9. doi: 10.1016/j.rmed.2006.03.012. Epub 2006 May 2. PMID 16650970
- [Result] McShane PJ, Naureckas ET, Tino G, Strek ME. Non-cystic fibrosis bronchiectasis. Am J Respir Crit Care Med. 2013 Sep 15;188(6):647-56. doi: 10.1164/rccm.201303-0411CI. PMID 23898922
- [Result] Flume PA, Chalmers JD, Olivier KN. Advances in bronchiectasis: endotyping, genetics, microbiome, and disease heterogeneity. Lancet. 2018 Sep 8;392(10150):880-890. doi: 10.1016/S0140-6736(18)31767-7. PMID 30215383
- [Result] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110